CLINICAL TRIAL: NCT03566901
Title: Robot-assisted Locomotor and Stair Climbing Training for Improving Mobility and Participation in Daily Activities in Persons Affected by Stroke: a Multicenter Randomized Controlled Clinical Trial
Brief Title: Robot-Assisted Stair Climbing Training
Acronym: RASCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Collaborators: Marialuisa Gandolfi (Unknown); Christian Geroin (Unknown); Eleonora Dimitrova (Unknown); Nicola Valè (Unknown)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Professor of Rehabilitation Medicine, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STAIRs Trial
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Stroke
Keywords: Balance, Gait, Rehabilitation, Stroke, Robotics, Postural
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A multisite single blind randomized controlled trial involving the 3 clinical sites (Verona, Bolzano, Monza) will be performed, according to the CONSORT Statement (www.consort-statement.org). The PIs will be responsible for the randomization procedures. If eligible, patients will be randomly allocated (allocation ratio 1:1) to the experimental (EG) or conventional physiotherapy (CP) using computer-generated random numbers (www.randomization.com). In each site, one examiner blinded to group assignment will be responsible for assessments.
  Prior to the start of the study the EG and CP protocols will be designed. To ensure uniformity in the delivery of treatments, one therapist from each center will be taught to training protocols by the research collaborators. Participants will receive 50-min, individual treatment sessions as outpatients 2 days a week for 5 consecutive weeks, for a total of 10 sessions. For each Unit one physiotherapist will be assigned to the EG and one to the CP.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-Assisted Stair Climbing Training (Experimental): Each session will consist of the G-EO System training and stretching exercises. Total net treatment time/session: 50 minutes. Physiotherapists will alter constraints to grade tasks according to patient ability. The training complexity will be increased, as the patient will improve in performance (i.e. increasing gait speed, reducing body weight support, increasing the number of repetition). Heart rate during training sessions will be monitored using a Polar V800. Heart rate will not exceed the threshold of 120 bpm.
  Interventions: Device: G-EO System
- Conventional Physiotherapy (Active Comparator): 50 min of overground walking training and stair climbing up/down and lower limb mobilization and stretching exercise.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Device: G-EO System — The G-EO Systems can reproduce the gait pattern and realistically simulates the ability to carry out stairs up and stairs down. It provides real-time feedback on the patient's movements with the Visual Scenario and offers the possibility to experience augmented reality further enhance the effectiveness of each therapy session. An intelligent control (G-EO System Evolution) reacts and adapts to each patient's individual capability by either supporting the patient - active assistive mode - or increasing resistance - active mode. The G-EO Systems rehabilitation robot allows to secure the subjects with a harness while they stood on the foot plates of the machine. The foot plates has 3 DoF each, allowing to control the length and the height of the steps and the foot plate angles. The maximum step length corresponded to 550 mm, the maximum achievable height of the steps is 400 mm, the maximum angles is ±90°. The maximum speed of the foot plates is 2,3 km/h.
  Arms: Robot-Assisted Stair Climbing Training
Other: Conventional Physiotherapy — Overground walking training including real stair climbing up/down and lower limb mobilization and stretching exercises.
  Arms: Conventional Physiotherapy

SUMMARY:
Stair climbing up and down is an essential part of everyday's mobility. Physiotherapy is focused on muscle strengthening, real floor walking and stairs climbing tasks, but these methods do not stress in terms of intensity stair-climbing practice. The aims of this study is to compare whether an intensive robot-assisted stair climbing training (RASCT) is more effective than conventional physiotherapy (CP) for improving stair climbing ability, gait and postural control in stroke patients.

DETAILED DESCRIPTION:
Trial design: A pilot randomized (allocation ratio 1:1), single blind clinical trial (RCT) comparing the effects between the experimental [Robot-Assisted Stair Climbing Training group (RASCT)] and control group (Conventional Physiotherapy, CP) in improving stair climbing ability and postural control in stroke patients. The examiner will be blind to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic or hemorrhagic stroke;
* More than or equal to 3 months post stroke;
* Age>18 years;
* Mini- Mental State Examination (MMSE) score more than 23;
* Ability to stand for at least 1 min without arm support; ability to walk independently for at least 10 m with or without walking aids;
* Functional Ambulation Category score equal or more than 1.
* Signed informed consent form

Exclusion Criteria:

* Severe cognitive or communicative disorders that hamper collaboration;
* Unstable cardiovascular system conditions (i.e. labile compensated cardiac insufficiency, angina pectoris), deep vein thrombosis, severe neurological or orthopedic diseases which massively affect lower limb mobility; severe joint misalignment;
* Treatment of lower limb spasticity (i.e. botulinum toxin) in the 3 months prior to the start of the study and/or during its execution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
The time required to climb Up and Down 9 stairs (seconds) | 1 day
  (seconds)

SECONDARY OUTCOMES:
6-Minute Walking Test evaluates walking endurance. | 1 day
  (meters)
The 10-Meter Walking Test evaluates gait speed. | 1 day
  (seconds)
The Berg Balance Scale evaluates standing balance during functional activities. | 1 day
  (score)
The Timed Up and Go test evaluates person's mobility. | 1 day
  (seconds)
The Modified Ashworth Scale evaluates muscle spasticity. | 1 day
  (score)
Fatigue Severity Scale | 1 day
  (score)
Number of steps performed with the Robot and without. | 1 day
  (number of steps)
Borg Scale | 1 day
  (score)
Functional Ambulation Category (FAC); | 1 day
  (score)
Dynamic Gait Index (DGI) | 1 day
  (score)
Barthel Index | 1 day
  (score)
European Stroke Scale | 1 day
  (score)
EMG gait | 1 day
  (phases of muscles activation)
Stabilometric assessment | 1 day
  (center of pressure parameters)
Blood pressure | 1 day
  mmg
heart beat | 1 day
  (number per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania, MD, Prof, Principal Investigator — Universita di Verona
Locations (2):
- Italy (2):
  - University of Verona, Verona
  - UOC Neurorehabilitation, Verona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Morone G, Paolucci S, Cherubini A, De Angelis D, Venturiero V, Coiro P, Iosa M. Robot-assisted gait training for stroke patients: current state of the art and perspectives of robotics. Neuropsychiatr Dis Treat. 2017 May 15;13:1303-1311. doi: 10.2147/NDT.S114102. eCollection 2017. PMID 28553117
- [Derived] Gandolfi M, Vale N, Dimitrova E, Zanolin ME, Mattiuz N, Battistuzzi E, Beccari M, Geroin C, Picelli A, Waldner A, Smania N. Robot-Assisted Stair Climbing Training on Postural Control and Sensory Integration Processes in Chronic Post-stroke Patients: A Randomized Controlled Clinical Trial. Front Neurosci. 2019 Oct 24;13:1143. doi: 10.3389/fnins.2019.01143. eCollection 2019. PMID 31708735